CLINICAL TRIAL: NCT06755567
Title: Application of MRI Radiomics Features in Neoadjuvant Therapy of Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1175-02
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer; Neoadjuvant Therapy; Immunotherapy; Chemotherapy; Pathologic Complete Response
MeSH Terms: conditions — Head and Neck Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HNSCC with NACI: HNSCC with neoadjuvant chemoimmunotherapy, following by radical sugery.
  Interventions: Diagnostic Test: MRI-based radiomics-clinical model

INTERVENTIONS:
Diagnostic Test: MRI-based radiomics-clinical model — Response to NACI was predicted using MRI-based radiomics-clinical model.

SUMMARY:
Head and neck squamous cell carcinoma is the sixth most common malignant tumor in the world. Neoadjuvant therapy, including neoadjuvant chemotherapy and immunotherapy, is recommended for patients with locally advanced head and neck cancer. The response to neoadjuvant therapy varies among the patients. It is reported that about 37% of the patients achieve pathological complete response after receiving neoadjuvant therapy, who would achieve a better prognosis compared with the patients with non-pathological complete response. It is significant to predict and assess response to neoadjuvant therapy for the patients with head and neck cancer accurately, which could assist in formulating individualized therapeutic regimens. MRI has good soft tissue resolution and is a common preoperative examination method. However, this method lacks the ability to accurately predict the probability of patients achieving pathological remission after neoadjuvant therapy. At present, it is a novel and effective method to construct a model to predict the efficacy of neoadjuvant therapy based on MRI image omics analysis, and certain achievements have been made in breast cancer and rectal cancer. In this study, multi-sequence MRI was combined with clinical risk factors to construct an imaging omics model to predict the probability of pathological complete remission of patients with head and neck squamous cell carcinoma after neoadjuvant therapy, and to accurately identify diagnostic imaging remission, so as to better assist clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* (a) patients pathologically diagnosed as head and neck squamous cell carcinoma;
* (b) patients receiving two or three courses of neoadjuvant therapy (traditional chemotherapy plus PD-1 inhibitor);
* (c) MR scan within 30 days before the first course of neoadjuvant therapy;
* (d) patients undergoing radical surgical dissection following neoadjuvant therapy;
* (e) complete clinical data available.

Exclusion Criteria:

* (a) previous head and neck treatment history;
* (b) obvious motion or metal artifacts on the MRI image;
* (c) distant metastasis;
* (d) concurrent malignancies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck squamous cell carcinoma, who were treated in Sun Yat-sen Memorial Hospital between January 2020 and October 2023, were included and randomly allocated into a training set (n = 300) and an internal validation set (n = 150). Patients treated in Sun Yat-Sen University Cancer Centre, Shenshan Medical Centre, Memorial Hospital of Sun Yat-sen University and Huizhou First Hospital between January 2020 and April 2024, were assigned as an external validation set (n = 150) . Patients treated in Sun Yat-sen Memorial Hospital, Sun Yat-Sen University Cancer Centre, Shenshan Medical Centre, Memorial Hospital of Sun Yat-sen University and Huizhou First Hospital between October 2024 and June 2025, were assigned as an prospective validation set (n = 150) .
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the area under the receiver operating characteristic (AUROC) curves | 2021.1-2023.2